CLINICAL TRIAL: NCT01265615
Title: Phase 4 Study of Paricalcitol and Calcitriol for Reparative Management of Chronic Allograft Dysfunction and Renocardiac Syndrome in Vitamin D Insufficient Renal Transplant Recipients
Brief Title: Paricalcitol Versus Calcitriol for the Management of Renocardiac Syndrome in Renal Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ural State Medical University (Other)
Collaborators: Ural Institute of Cardiology (Other); De Haar Research Foundation (Other)
Responsible Party: Principal Investigator, Alexander Kharlamov, Lecturer at the Ural Medical University, Ural State Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VDCRS03
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Cardiorenal Syndrome; Chronic Allograft Nephropathy
Keywords: chronic allograft nephropathy; stem-progenitor cells; cardiorenal syndrome; calcitriol; paricalcitol; cholecalciferol; cardiac repair; renal repair
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — paricalcitol; Calcitriol; Cholecalciferol; Alendronate; Dietary Supplements; Diet; Solar System; Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Paricalcitol treatment (Active Comparator): 6-8 μg daily per os (orally) without special diet
  Interventions: Drug: Paricalcitol
- Calcitriol treatment (Active Comparator): 2-4 μg daily orally under with dietary restrictions of vitamin D
  Interventions: Drug: Calcitriol
- Cholecalciferol (Active Comparator): alendronate sodium/ cholecalciferol capsules with recommended daily allowance equals 1200-2400 IU per day
  Interventions: Drug: Cholecalciferol
- Supplemental (Other): intake of cholecalciferol in food and multivitamins, less than 400-900 IU per day
  Interventions: Dietary Supplement: Supplemental

INTERVENTIONS:
Drug: Paricalcitol — paricalcitol group (6-8 μg daily per os - orally - without special diet)
  Other Names: Zemplar
  Arms: Paricalcitol treatment
Drug: Calcitriol — calcitriol group (2-4 μg daily orally under with dietary restrictions of vitamin D)
  Other Names: Rocaltrol
  Arms: Calcitriol treatment
Drug: Cholecalciferol — cholecalciferol group (intake of cholecalciferol with recommended daily allowance equals 1200-2400 IU per day)
  Other Names: Fosamax
  Arms: Cholecalciferol
Dietary Supplement: Supplemental — intake of cholecalciferol in food and multivitamins, less than 400-900 IU per day
  Other Names: Diet, sun, multivitamin drugs, food
  Arms: Supplemental

SUMMARY:
We hypothesize that paricalcitol and calcitriol in dose-dependent manner are effective for the management of chronic allograft dysfunction (CAD), protection and repair of kidney and heart, management of chronic renocardiac syndrome (CRS). We assume that paricalcitol can have some advantages if compare with calcitriol or cholecalciferol due to absence of calcemic and phosphatemic complications alongside with great beneficial potential.

DETAILED DESCRIPTION:
Paricalcitol and calcitriol are identically effective for the management of chronic allograft dysfunction (CAD), protection and repair of kidney and heart, management of chronic renocardiac syndrome (CRS). Vitamin D can reduce progression of CAD. Activation of VDR in proximal part of nephron leads to rapid non-genomic beneficial effects with urgent multilevel protection of the most functionally important portion of kidney. Rising expression of VDR in distal portions of nephron stimulates slows genomic effects with some local repair responses.

Hormone D may stimulate recruitment and activity of the different origin stem-progenitor cells (SPCs) with beneficial effects on different stages of regeneration by force of para- and autocrine activity. SPCs are revealing mostly in interstitium and among fibroblast-like cells. Vitamin D did not confirm efficacy as a tool for management of mesenchymal stem cells (MSCs) in human however it needs more research experimental evidences due to multifactorial influence on SPCs in human being including immunosuppressive and bone-marrow-related effects of cyclosporine in kidney transplant (Tx) patients. Paricalcitol and calcitriol can slow down migration and infiltration of MSC into interstitium and vessel wall. The side population of mature and SPCs (first of all, with bone-marrow and mesenchymal phenotype) is the most metabolically and functionally active portion of cells with high sensitivity to vitamin D receptor (VDR) activation that responsible for repair of tissue.

The most optimal scheme of treatment with vitamin D in patients with CAD and CRS is an administration of paricalcitol with dose 2-4 μg daily and supplemental intake of vitamin D including special diet, multivitamins, and others with optimal dose until 1800 international units (IU) but excluding insolation as a factor of skin carcinoma. High-dose medicinal intake of calcitriol (until 6 mcg and higher) showed relatively high efficacy but rather excessive level of complications mediated with mineral metabolism.

Paricalcitol and calcitriol may significantly improve contractility of myocardium and reduce cardiovascular risk, heart failure (HF) and hypertension with some beneficial effects on cardiorenal axis and renin-angiotensin-aldosterone system.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75
* Male
* History of chronic kidney disease and cardiorenal syndrome
* Written informed consent

Exclusion Criteria:

* Female
* Acute illness
* Life-threat competitive illness
* Mental disorders
* Endocrinologic diseases (including diabetes mellitus, hyperparathyroidism, and other thyroid disorders)
* Need for dialyses
* Hypercalcemia
* Concomitant use of hormone or cytokine medication
* Participation to any drug-investigation during the previous 60 days as checked with VIP check

Ages: 40 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-10; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kharlamov, M.D., Principal Investigator — Ural Institute of Cardiology; Alexander Perrish, M.D., Principal Investigator — Ural State Medical University
Locations (2):
- De Haar Research Foundation, Rotterdam, South Holland, Netherlands
- Ural Institute of Cardiology, Yekaterinburg, Russia

REFERENCES:
- [Result] Kharlamov AN, Perrish AN, Gabiskii IaL, Ronne Kh, Ivanova EIu. [Vitamin D in the treatment of cardiorenal syndrome in patients with chronic nephropathy]. Kardiologiia. 2012;52(3):33-44. Russian. PMID 22839442
- See also: Ural Institute of Cardiology — http://www.cardio-burg.ru

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 120 patients (Russian and dutch caucasian, kidney recipients with vitamin D deficiency defined as 25(OH)D < 30 ng/mL) were assigned on the basis of Ural Institute of Cardiology. Nine of the 120 patients were subsequently excluded due to protocol violation. All the patients had given their written informed consents.
Groups:
- Paricalcitol Treatment: 6-8 μg daily per os without special diet
Period: Overall Study
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Started | 30 | 30 | 30 | 30
Completed | 28 | 28 | 26 | 27
Not Completed | 2 | 2 | 4 | 3
Not completed — Protocol Violation | 2 | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 28 | 26 | 27 | 109
  >=65 years | 2 | 2 | 4 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (4) | 59 (4) | 58 (5) | 57 (4) | 58 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 30 | 30 | 30 | 30 | 120
Region of Enrollment [Number; unit: participants]
  Russian Federation | 30 | 30 | 30 | 30 | 120

OUTCOME MEASURES:

1. Primary Outcome: CAD (Chronic Allograft Dysfunction) Degree
Description: Beyond 180 days, chronic allograft dysfunction (CAD) was characterized by mean Banff degree (revised 2005/2007 criteria) with the data of renal biopsy material. Renal tissue was recovered during routined biopsy. We assessed antibody-mediated rejection, borderline changes, T-cell-mediated rejection, interstitial fibrosis and tubular atropthy, and other changes. Grades:
  Grade I. Mild interstitial fibrosis and tubular atrophy (<25% of cortical area) II. Moderate (26-50%) III. Severe (>50%) (may include non-specific vascular and glomerular sclerosis)
Time Frame: day 180 after Tx (transplantation)
Measure: Mean (Standard Deviation); unit: Scores on a Banff scale
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
Scores on a Banff scale | 1.24 (0.14) | 1.22 (0.42) | 1.43 (0.22) | 1.68 (0.36)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Heart Failure (HF)
Description: NYHA (New York Heart Association) functional class verified with veloergometry probe and by NYHA clinical classification NYHA Class Symptoms I No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  II Mild symptoms and slight limitation during ordinary activity. III Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).
  Comfortable only at rest. IV Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
Time Frame: on day 180 after Tx (transplantation)
Population: A total of 120 patients (Russian and dutch caucasian, kidney recipients with vitamin D deficiency defined as 25(OH)D < 40 nmol/l) were assigned. Analysis was per protocol.
Measure: Mean (Standard Deviation); unit: NYHA functional class of HF
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
NYHA functional class of HF | 1.8 (0.2) | 1.9 (0.3) | 1.9 (0.1) | 2.5 (0.2)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

3. Secondary Outcome: GFR (Glomerular Filtration Rate)
Description: Estimated glomerular filtration rate (eGFR) was calculated using the abbreviated form of the Modification of Diet in Renal Disease (MDRD) study equation: eGFR = exp (5.228 - 1.154 × ln (serum creatinine) - 0.203 × ln (age). Concerning of GFR with Tc99m DTPA renography was used for the complex analysis of renal function. Camera based GFR estimated from Tc99m DTPA renography was named Gates GFR.
Time Frame: on day 180
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
ml/min/1.73 m^2 | 84 (11) | 81 (9) | 76 (10) | 54 (9)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

4. Secondary Outcome: CAD (Chronic Allograft Dysfunction) Degree
Description: CAD degree measured by Banff score after routine renal biopsy (revised 2005/2007 criteria). We assessed antibody-mediated rejection, borderline changes, T-cell-mediated rejection, interstitial fibrosis and tubular atropthy, and other changes. Grades:
  Grade I. Mild interstitial fibrosis and tubular atrophy (<25% of cortical area) II. Moderate (26-50%) III. Severe (>50%) (may include non-specific vascular and glomerular sclerosis)
Time Frame: on day 90
Measure: Mean (Standard Deviation); unit: Scores on a Banff scale
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
Scores on a Banff scale | 1.24 (0.14) | 1.22 (0.42) | 1.43 (0.22) | 1.68 (0.36)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

5. Secondary Outcome: Serum Creatinine
Description: After an overnight fast, plasma concentrations of hemoglobin, creatinine, cholesterol, glucose, total calcium, and phosphate were measured using an autoanalyzer as described by Adorini L. (2005)
Time Frame: on day 180 after Tx
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
mg/dL | 2.5 (0.9) | 2.5 (0.7) | 2.8 (0.7) | 4.1 (1.1)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

6. Secondary Outcome: Number of Circulating SP (Side Population) Stem-Progenitor Cells
Description: Renal cells and solid tissue were obtained from the normal portion of cortex obtained from surgically removed kidneys or by standart biopsy on day 180. Cytofluorimetric analysis and immunofluorescence were performed as described by Oliver J.A. (2004). Sorting and analysis of different cells was done on a FACS (fluorescent activated cell sorting) and by flow cytometry. Cells were analyzed with EPICS systems (Beckman Coulter). Quantification of mRNA expression was achieved using Assays-on-Demand gene expression kits and the ABI PRISM 7000 Sequence Detection System (Applied Biosystem).
Time Frame: on day 180
Measure: Mean (Standard Deviation); unit: per cent of SP cells
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
per cent of SP cells | 7.6 (0.9) | 6.5 (1) | 5.7 (0.8) | 4.2 (0.7)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

7. Secondary Outcome: VDR (Vitamin D Receptor) Expression in Myocardium
Description: VDR content was determined by using an ELISA developed in this laboratory. The protein concentration of the homogenates was determined by the method of Bradford (1976), using BSA as a standard.
Time Frame: on day 180
Measure: Mean (Standard Deviation); unit: fmol VDR/ mg protein
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
fmol VDR/ mg protein | 801 (112) | 715 (96) | 654 (88) | 389 (77)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

8. Secondary Outcome: VDR (Vitamin D Receptor) Expression in Kidney
Description: as for outcome 7
Time Frame: on day 180
Measure: Mean (Standard Deviation); unit: fmol VDR/ mg protein
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
fmol VDR/ mg protein | 584 (103) | 599 (102) | 478 (79) | 333 (62)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

9. Secondary Outcome: Systolic Blood Pressure
Description: SBP measured by routine method
Time Frame: on day 180
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
mmHg | 143 (22) | 141 (9) | 147 (13) | 165 (19)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

10. Secondary Outcome: Coronary Calcium Score
Description: Bone mineral density assessed by dual-energy X-ray absorptiometry (DXA) of the whole body, lumbar spine and hip was performed using Hologic scanners (QDR 1000W or QDR 2000). The total Agatston coronary calcium score (CCS) was measured as the sum of calcified plaque scores of all the coronary arteries. The amount of calcium present in the coronary arteries is scored according to the Agatson scale, as follows: 0 - no identifiable disease; 1 to 99 - mild disease; 100 to 399 - moderate disease; 400 or higher - severe disease.
Time Frame: on day 180
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Number analyzed (Participants) | 28 | 28 | 26 | 27
units on a scale | 530 (423) | 611 (502) | 524 (122) | 990 (120)
Statistical Analysis 1: Comparison: Paricalcitol Treatment vs Calcitriol Treatment vs Cholecalciferol vs Supplemental; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Paricalcitol Treatment | Calcitriol Treatment | Cholecalciferol | Supplemental
Serious Adverse Events (participants affected / at risk) | 9/30 | 21/30 | 6/30 | 8/30
Other Adverse Events (participants affected / at risk) | 10/30 | 15/30 | 9/30 | 9/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol Treatment (N=30) | Calcitriol Treatment (N=30) | Cholecalciferol (N=30) | Supplemental (N=30)
Hypercalcemia (Endocrine disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypophospatemia (Endocrine disorders) | 7 (7) | 16 (16) | 5 (5) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paricalcitol Treatment (N=30) | Calcitriol Treatment (N=30) | Cholecalciferol (N=30) | Supplemental (N=30)
Pain (General disorders) | 4 (4) | 4 (4) | 5 (5) | 4 (4)
Fatigue (General disorders) | 5 (5) | 7 (7) | 3 (3) | 4 (4)
Viral Infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Allergic Infection (Immune system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Back Pain (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
General Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3)
Fever (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Infection Fungal (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Conjuctivitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decreased libido (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Increased hypertension (Cardiac disorders) | 4 (4) | 3 (3) | 5 (5) | 6 (6)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrhythmias (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Anorexia (Psychiatric disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 5 (5) | 4 (4) | 7 (7)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1)
Taste perversions (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2) | 2 (2) — Predominantly metallic taste
Polydipsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Edema (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 5 (5) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Leg Cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2) | 4 (4)
Vertigo (Nervous system disorders) | 3 (3) | 2 (2) | 4 (4) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 3 (3)
Increased Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No